CLINICAL TRIAL: NCT00982605
Title: EBUS-guided TBNA for Molecular Diagnostic of Mediastinal Lymph Nodes
Brief Title: EBUS-guided TBNA for Molecular Diagnostic of Mediastinal Lymph Nodes (LN)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Felix Herth, Thoraxklinik Heidelberg
Other Study IDs: MK01
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lymph nodes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- non small cell lung cancer: cancer patients
  Interventions: Procedure: EBUS_TBNA

INTERVENTIONS:
Procedure: EBUS_TBNA — EBUS during bronchoscopy
  Other Names: EBUS-TBNA scope, Olympus Medical

SUMMARY:
The purpose of this study is to perform molecular diagnostic in mediastinal lymph nodes of non-small cell lung cancer patients sampled by endobronchial ultrasound guided finde needle aspiration (EBUS-TBNA).

DETAILED DESCRIPTION:
NSCLC is a common cancer. Accurate and early staging has a significant impact on outcome. EBUS-TBNA of involved mediastinal lymph nodes is critical. Molecular markers could improve mediastinal staging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Samples are collected before surgery or before any therapy
* ECOG 0 or 1
* Clinical stage I-II, T1-2, N0-1, M0)
* Surgically respectable
* Patient with enlarged med. lymphnodes (control group)

Exclusion Criteria:

* Previous RT/CHT
* Previous or current cancer of other entity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with operable non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Estimated); Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kreuter, MD, Study Director — Thoraxklinik Heidelberg, Germany
Locations (1):
- Thoraxklinik Heidelberg, Dept. of Pneumology and Respiratory Critical care, Heidelberg, Germany

REFERENCES:
- [Background] Herth FJ, Annema JT, Eberhardt R, Yasufuku K, Ernst A, Krasnik M, Rintoul RC. Endobronchial ultrasound with transbronchial needle aspiration for restaging the mediastinum in lung cancer. J Clin Oncol. 2008 Jul 10;26(20):3346-50. doi: 10.1200/JCO.2007.14.9229. Epub 2008 Jun 2. PMID 18519953
- [Background] Herth FJ, Eberhardt R. Actual role of endobronchial ultrasound (EBUS). Eur Radiol. 2007 Jul;17(7):1806-12. doi: 10.1007/s00330-006-0497-6. Epub 2007 Jan 6. PMID 17206430
- [Background] Herth FJ, Ernst A, Eberhardt R, Vilmann P, Dienemann H, Krasnik M. Endobronchial ultrasound-guided transbronchial needle aspiration of lymph nodes in the radiologically normal mediastinum. Eur Respir J. 2006 Nov;28(5):910-4. doi: 10.1183/09031936.06.00124905. Epub 2006 Jun 28. PMID 16807262
- [Background] Herth FJ, Eberhardt R, Vilmann P, Krasnik M, Ernst A. Real-time endobronchial ultrasound guided transbronchial needle aspiration for sampling mediastinal lymph nodes. Thorax. 2006 Sep;61(9):795-8. doi: 10.1136/thx.2005.047829. Epub 2006 May 31. PMID 16738038
- [Background] Al-Haddad M, Wallace MB. Molecular diagnostics of non-small cell lung cancer using mediastinal lymph nodes sampled by endoscopic ultrasound-guided needle aspiration. Cytopathology. 2006 Feb;17(1):3-9. doi: 10.1111/j.1365-2303.2006.00318.x. PMID 16417559